CLINICAL TRIAL: NCT03540043
Title: 4-Week Multicenter, Randomized, Double-Blind, Parallel-Group, Vehicle-Controlled Safety and Efficacy Study of PUR 0110 (Thykamine™) Cream Applied Twice Daily in Mild-to-Moderate Atopic Dermatitis
Brief Title: Thykamine Safety and Efficacy Study in Mild-to-Moderate Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PurGenesis Technologies Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DV16-PUR0110-C001
Record Dates: First submitted 2018-04-15; First posted 2018-05-30 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2020-06

CONDITIONS: Atopic Dermatitis Eczema
Keywords: Mild moderate atopic dermatitis

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind, Parallel-Group, Placebo-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Treatment were packaged in identical jars. Eligible patients will be randomized in a 1:1:1:1 ratio to receive either one of 3 concentrations of PUR 0110 cream (0.05%, 0.1% and 0.25%) or vehicle (placebo).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Placebo (Placebo Comparator): Administration of Placebo
  Interventions: Drug: Administration of Placebo
- PUR0110 (Thykamine) 0.05% (Experimental): Administration of PUR0110 (Thykamine) 0.05%
  Interventions: Drug: Administration of PUR0110 (Thykamine) 0.05%
- PUR0110 (Thykamine) 0.10% (Experimental): Administration of PUR0110 (Thykamine) 0.10%
  Interventions: Drug: Administration of PUR0110 (Thykamine) 0.1%
- PUR0110 (Thykamine) 0.25% (Experimental): Administration of PUR0110 (Thykamine) 0.25%
  Interventions: Drug: Administration of PUR0110 (Thykamine) 0.25%

INTERVENTIONS:
Drug: Administration of Placebo — Botanical Drug Phase 2 clinical study
  Other Names: Placebo control
  Arms: Placebo
Drug: Administration of PUR0110 (Thykamine) 0.05% — Botanical Drug Phase 2 clinical study
  Other Names: Active arm
  Arms: PUR0110 (Thykamine) 0.05%
Drug: Administration of PUR0110 (Thykamine) 0.1% — Botanical Drug Phase 2 clinical study
  Other Names: Active arm
  Arms: PUR0110 (Thykamine) 0.10%
Drug: Administration of PUR0110 (Thykamine) 0.25% — Botanical Drug Phase 2 clinical study
  Other Names: Active arm
  Arms: PUR0110 (Thykamine) 0.25%

SUMMARY:
A Phase 2, multicenter, double-blind, placebo control study evaluating the safety and efficacy of Thykamine in adult patient suffering of mild-to-moderate Atopic Dermatitis

DETAILED DESCRIPTION:
4-week Multicenter, Randomized, Double-Blind, Parallel-Group, Vehicle-Controlled Safety and Efficacy Study of Three Concentrations (0.05%, 0.1% and 0.25%) of PUR 0110 (Thykamine™) Cream Applied Twice Daily in Mild-to-Moderate Atopic Dermatitis.

ELIGIBILITY:
Inclusion criteria

The patient must meet all the following criteria to be enrolled in the study:

1. Male or female patients, aged 18 years or older at the screening visit.
2. Patients with diagnosis of AD for at least 6 months prior to Day 0 visit as defined by the criteria of Hanifin and Rajka (Acta Derm Venereol. 1980).
3. Patients with BSA ≥ 1 % and ≤ 15% at Day 0 (excluding palms, soles and scalp).
4. Patients with IGA score of 2 to 3 (mild-to-moderate) at Day 0.
5. Female patients of childbearing potential must have a negative pregnancy test (serum Beta-hCG) at the screening visit - unless they are surgically sterile (hysterectomy, bilateral oophorectomy or tubal ligation), in a menopausal state for at least a year, clinically diagnosed infertile, or have a same-sex partner or are abstinent.
6. In addition, females of childbearing potential or a male patient with a female partner must be willing to use an effective contraceptive method for at least 30 days (12 weeks for hormonal contraceptives) before Day 0 and at least 1 month after the last study drug administration. Effective contraceptive methods include:

   * Barrier methods such as condom, sponge or diaphragm combined with spermicide in foam, gel or cream;
   * Hormonal contraception (oral, intramuscular, implant or transdermal) which include Depo Provera, Evra and Nuvaring; and
   * Intrauterine device (IUD).
7. Patients must be capable of giving informed consent and the consent must be obtained prior to any study related procedures.

Exclusion criteria

1. Patient with BSA > 15% (excluding palms, soles and scalp).
2. Female who is pregnant or lactating or wishes to become pregnant during the study period.
3. Patient with a history of any confounding inflammatory skin diseases or any other skin disease, e.g., psoriasis, rosacea, erythroderma or ichthyosis, that could impair his/her safety during the study or interfere with the evaluation of AD.
4. Patient with spontaneously improving or rapidly deteriorating AD.
5. Patient with active allergic contact dermatitis or other non-atopic forms of dermatitis.
6. Patient with active cutaneous bacterial or viral or fungal infection in any treatment area at baseline (e.g., clinically infected AD).
7. Patient with acute infections.
8. Patient with a history or presence of Netherton's syndrome, immunological deficiencies or diseases, diabetes, malignancy, psychological disorders, serious active or recurrent infection, clinically significant severe renal insufficiency or severe hepatic disorders - which might cause this study to be detrimental to the patient or that may confound the study results or interfere significantly with the patient's participation in the study.
9. Patient with bleeding disorders.
10. Patient with known seropositivity for the human immunodeficiency virus or evidence of active hepatitis B or C.
11. Patient has an unstable or serious medical condition, as defined by the investigator, which might cause this study to be detrimental to the patient or that may confound the study results or interfere significantly with the patient's participation in the study.
12. Patient has a history of alcoholism or drug abuse within 12 months prior to Day 0.
13. Patient with known allergy, or history of allergic reaction, or hypersensitivity to spinach, spinach tablet, spinach powder or spinach extract; to mushrooms; or any ingredients present in PUR 0110.
14. Patient with a history of severe food allergies.
15. Patient with sunburn, extensive scarring, or pigmented lesion(s) in any treatment area at baseline (Day 0), which would interfere with evaluations.
16. Use within 4 weeks prior to baseline (Day 0) of oral or intravenous corticosteroids, UVA/UVB therapy, PUVA (psoralen plus ultraviolet A) therapy, tanning booths, non-prescription UV light sources, immunomodulators or immunosuppressive therapies, interferon, or cytotoxic drugs.
17. Use within 2 weeks of baseline (Day 0) of systemic antibiotics, calcipotriene or other vitamin D preparations, or retinoids.
18. Use within 2 weeks of baseline (Day 0) of oral natural health products or vitamins containing lutein.
19. Use within 1 week prior to baseline (Day 0) of antihistamines, topical antibiotics, topical corticosteroids, topical calcineurin inhibitors or other topical drug products used for treating AD. Inhaled corticosteroids for stable medical conditions are allowed.
20. Use within 24 hours prior to baseline (Day 0) of any topical product (e.g., sunscreens, lotions, creams) in the areas to be treated, except for bland emollient (moisturizer).
21. Use of an investigational agent within 4 weeks or 5 half-lives prior to Day 0 (whichever is longer).
22. Patient not willing to minimize or avoid natural and artificial sunlight exposure during treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2017-10-23 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-06-03 (Actual)

PRIMARY OUTCOMES:
Efficacy as per investigator global assessment (IGA) | Baseline and 4 weeks
  Efficacy as per investigator global assessment (IGA) of clear (0), almost clear (1) at Day 29 and with a decrease from baseline in IGA of at least 2 grades at Day 29.

SECONDARY OUTCOMES:
Incidence and severity of adverse events (AEs) (systemic and local) | Baseline and 4 weeks
  Incidence and severity of adverse events (AEs) (systemic and local) as a measure of safety and tolerability of treatment for up to Day 29.
Change from baseline in Atopic Dermatitis (AD) score | Baseline and 4 weeks
  Change from baseline to Day 29 in the 4 individual signs/symptoms score of AD including: erythema, induration/papulation, excoriation and lichenification measured in the target lesion on a 4-point scale defined as : 0 = None; 1=Mild; 2=Moderate and 3=Severe
Change in pruritus | Baseline and 4 weeks
  Change from baseline to Day 29 in pruritus, measured on a 4-point scale defined as : 0=None; 1=Mild; 2=Moderate and 3=Severe
Proportion of patients with change in Investigator Global Assessment (IGA) | Baseline and 3 weeks
  • Proportion of patients with an IGA of clear (0), almost clear (1) and with a decrease from baseline in IGA of at least 2 grades at intermediate visits (Days 7, 14 and 21). Scores being defined as : 0=Clear ; 1=Almost Clear; 2:=Mild disease; 3=Moderate disease and 4 = Severe disease
Change in Eczema Area and Severity Index (EASI) | Baseline and 4 weeks
  Change from baseline to Day 29 in Eczema Area and Severity Index (EASI).Four body regions are considered separately and include: Head and neck; Trunk ; Upper extremities; Lower extremities (including the buttocks).Extent of Eczema in these regions is being scored as follow : 0 = 0% involvement; 1= 1-9%; 2 = 10-29%; 3= 30-49%; 4= 50-69%; 5= 70-89% and 6= 90-100%. Severity of erythema, edema/papulation, excoriation and lichenification , for each region is scaled as : 0=none; 1= mild; 2= moderate and 3= severe. Final EASI score is the sum of the 4 region scores and ranges from 0-72.

OTHER OUTCOMES:
EASI improvement | Baseline and 4 weeks
  Proportion of patients with at least a 50% and 75% improvement in EASI (EASI50) at Day 29 as compared to baseline
Change from baseline in body surface area (BSA). | Baseline and 4 weeks
  Change from baseline to Day 29 in body surface area (BSA) affected by disease.
Change from baseline in Dermatology Life Quality Index (DLQI). | Baseline and 4 weeks
  Change from baseline to Day 29 in Dermatology Life Quality Index (DLQI) evaluating the impact on Quality of life scale : Very much ; A lot; a little or Not at all.
Change from baseline in Patient-Oriented Eczema Measure (POEM). | Baseline and 4 weeks
  Change from baseline to Day 29 in Patient-Oriented Eczema Measure (POEM) investigating the number of days patients have been subjected, due to eczema, to itchy skin, sleep disturbance; skin bleeding; skin weeping; skin craked; skin flaking and skin dryness. Scale defined as : 0 = no days; 1= 1-2 days; 2= 3-4 days; 3= 5-6 days; 4 = everyday

CONTACTS AND LOCATIONS:
Overall Officials: Yves Poulin, MD, Study Director — Centre de Recherche Dernatologique du Quebec; Wei Jing Loo, MD, Study Director — DermEffects
Locations (12):
- Canada (12):
  - SimcoDerm Medical and Surgical Dermatology Center, Barrie, Ontario
  - Manna Research Inc. (Burlington North), Burlington, Ontario
  - DermEffects, London, Ontario
  - Lynderm Research inc., Markham, Ontario
  - Manna Research Inc. (Toronto), Toronto, Ontario
  - Windsor Clinical Research Inc., Windsor, Ontario
  - DermEdge Research imc., Mississauga, Ontation
  - Q&T Research Chicoutimi, Chicoutimi, Quebec
  - Dr. Isabelle Delorme Inc., Drummondville, Quebec
  - Dr. David Gratton Dermatologue Inc., Montreal, Quebec
  - Centre de Recherche Saint-Louis, Québec, Quebec
  - Centre de Recherche Dermatologique du Quebec metropolitain (CRDQ), Québec

IPD SHARING:
Plan to Share IPD: No